CLINICAL TRIAL: NCT03071198
Title: Clinical Effect of Neoadjuvant Hierarchical Treatment Based on Chemotherapy for T3-4N0-2M0 Middle and Lower Rectal Cancer
Brief Title: Clinical Effect of Neoadjuvant Hierarchical Treatment Based on Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Binbin Cui, Director of colorectal surgery, Harbin Medical University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201702230001
Record Dates: First submitted 2017-02-26; First posted 2017-03-06 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Rectum Cancer
Keywords: Neoadjuvant Chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Intervention Model Description: This strategy is called "neoadjuvant hierarchical treatment" based on chemotherapy for rectal cancer. All patients with T3-4N0-2M0 middle and lower rectal caner will firstly receive neoadjuvant chemotherapy consisting of four cycles of XELOX. After four cycles, the patients achieved cCR or cPR will be perform the operation. And the patients who can not achieve cCR or cPR after the four cycles, then concurrent chemoradiotherapy will be added.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Preoperative neoadjuvant CT (Experimental): Give neoadjuvant chemotherapy for four cycle ,if achieve cCR or cPR after four cycles neoadjuvant chemotherapy , receive Total Mesorectal Excision(TME) ,then received the complete adjuvant therapy
  Interventions: Procedure: TME; Drug: neoadjuvant CT; Drug: adjuvant CT
- Preoperative neoadjuvant CT-RCT (Experimental): Give neoadjuvant chemotherapy for four cycle ,if not achieve cCR or cPR after four cycle neoadjuvant chemotherapy ,give concurrent chemo-radiotherapy,then additional neoadjuvant chemotherapy for 2 cycles ,then receive Total Mesorectal Excision(TME) ,then received the complete adjuvant therapy
  Interventions: Procedure: TME; Radiation: Concurrent chemo-radiotherapy; Drug: neoadjuvant CT; Drug: adjuvant CT
- Concurrent chemo-radiotherapy (Active Comparator): Give concurrent chemo-radiotherapy ,then receive Total Mesorectal Excision(TME) ,then received the complete adjuvant therapy
  Interventions: Procedure: TME; Radiation: Concurrent chemo-radiotherapy; Drug: adjuvant CT

INTERVENTIONS:
Procedure: TME — 1. Find the hypogastric nerve trunk in front of sacral promontory and protect it,be careful to use electrocautery hemostasis biased toward the side of rectal when handle lateral ligament of rectum and middle rectal artery and avoid to damage the pelvic plexus.
  2. At least a 2-cm margin to the lower edge of the tumor is adequate for distal bowel resection. Resect 5cm length distal rectal or all of the mesorectum.Check the integrity of the mesorectum in postoperative routine examination. Double stapling method is used for all low anastomosis operations.
Radiation: Concurrent chemo-radiotherapy — Three-dimensional conformal radiotherapy as following: CTV 44Gy/22 times＋GTV1 6Gy/3 times(2Gy/time/day，5 days a week，totally 5 weeks),if rectal tumors do not regress obviously, additional GTV2 is necessary, 5.4Gy/3 times (1.8Gy/time/day). At the same time, Capecitabine (850mg/m2, two times every day) will be taken on radiotherapy day
  Other Names: neoadjuvant RCT
  Arms: Concurrent chemo-radiotherapy; Preoperative neoadjuvant CT-RCT
Drug: neoadjuvant CT — CAPEOX protocol:Oxaliplatin 130mg/m2 ivgtt 2-6h dl;(Capecitabine 1000mg/m2 2 times a day lasts for 14 days Repeat every 3 weeks
  Other Names: neoadjuvant chemotherapy
  Arms: Preoperative neoadjuvant CT; Preoperative neoadjuvant CT-RCT
Drug: adjuvant CT — CAPEOX protocol:Oxaliplatin 130mg/m2 ivgtt 2-6h dl;(Capecitabine 1000mg/m2 2 times a day lasts for 14 days Repeat every 3 weeks
  Other Names: adjuvant chemotherapy

SUMMARY:
Clinical effect of neoadjuvant hierarchical treatment based on chemotherapy for T3-4N0-2M0 middle and lower rectal cancer

DETAILED DESCRIPTION:
By setting 3-Year disease-free survival (DFS) as main objective, the treatment strategy will be optimizing as neoadjuvant chemotherapy alone and chemo-radio-chemo sequential treatment.

ELIGIBILITY:
* Inclusion criteria
* Pathologically confirmed to be rectal adenocarcinoma.
* Distance < 10cm from the end of the tumor to the anal verge found on colonoscopy
* Tumor in stage T3-4N0-2 (pelvic MRI evaluation)
* Patients without distant metastases (such as liver and peritoneum, lungs, aortic lymph nodes)
* Patients with Karnofsky score greater ≥ 70
* WBC > 3.5 x 109/ml , PLT > 10 x 109/ml , TBIL<22.2 umol/l , BUN <7.14mmol/l , Cr<132umol/l or Ccr > 50ml/min (Evaluated using the Cockcroft-Gault formula: Creatinine clearance (male) = {(140 - age) x LBM (kg)} / {plasma creatinine (mg/dl) x 72} ; Creatinine clearance (female) = 0.85 x {(140 - age) x LBM(kg)}/ { plasma creatinine (mg/dl) x 72})
* Patients must sign the informed consent form
* Female subjects must be contraceptive during the trial
* Patients who did not receive any form of chemotherapy and radiotherapy
* No other important related diseases (such as other tumors, severe heart disease and central nervous system diseases, etc.)
* Age must be equal or more than 20 and must be equal or less than 70
* Exclusion criteria
* Previously received radiation therapy, chemotherapy or anti-tumor biological therapy
* Previously received immuno-suppressive therapy
* Participation in interventional clinical trial over the past time
* Suffering from malignant colonic neoplasms simultaneously
* With peripheral neuropathy(above WHO I level)
* Affected cognitive abilities because of neurological or psychiatric abnormalities Including central nervous system metastasis
* Medical history of severe allergies or allergic constitution
* Severe pulmonary or heart disease history
* Female patients who are in pregnancy or lactation and refuse contraception
* Previously with other malignant tumors
* Exit criteria
* Occurrence of bleeding, obstruction, perforation and other complications
* Occurrence of distant metastasis during the period of neoadjuvant therapy
* Adverse reactions, not be tolerated and do not want to continue to receive treatment
* Patients voluntarily quit
* Capecitabine-related Grade 4 Hand-Foot Syndrome

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | 3 years
  the treatment strategy will be optimizing as neoadjuvant chemotherapy alone and chemo-radio-chemo sequential treatment.

SECONDARY OUTCOMES:
Surgery related mortality and complication | 3 years
  Surgery related mortality and complication
Resection rate of R0 | 3 years
  Resection rate of R0
Pathologic complete remission (pCR) rate | 3 years
  Pathologic complete remission (pCR) rate
Tolerance after neoadjuvant treatment | 3 years
  Tolerance after neoadjuvant treatment
Predictor efficacy of neoadjuvant chemotherapy for DFS | 3 years
  Predictor efficacy of neoadjuvant chemotherapy for DFS

CONTACTS AND LOCATIONS:
Overall Officials: binbin cui, Principal Investigator — Harbin Medical University
Locations (1):
- Cancer Hospital Affiliated to Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided